CLINICAL TRIAL: NCT05362552
Title: The Positive Effects of an Urban Afforestation Activity on the Mental Health of Adults
Brief Title: Effects of Urban Afforestation Activity on Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Mármol, Associate Professor, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AfforestAffect
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: Green spaces; Nature-based activities; Urban afforestation; Horticultural therapy; Adults; Mental health; Affect; Vitality
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urban Afforestation Group (Experimental): Participants will perform an afforestation activity with a duration of 90 minutes.
  Interventions: Other: Urban Afforestation Program

INTERVENTIONS:
Other: Urban Afforestation Program — An afforestation program based on land cultivation and transplantation of several plants for 90 minutes will be implemented.
  Other Names: Nature-based activity; Afforestation activity

SUMMARY:
This single-group pretest-posttest clinical trial aims to evaluate the effects of a single-session afforestation activity on affect and vitality levels in a sample of young adults.

DETAILED DESCRIPTION:
The participants will perform an afforestation activity for a single session of 90 minutes. The therapists will direct the participants' attention to the visual, auditory, olfactory, and tactile features of the surrounding environment.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years.
* Any sex and gender.

Exclusion Criteria:

* Intake of any psychotropic medication.
* Other severe or medically unstable diseases that may interfere with participation.
* Severe cognitive impairment (Mini-Mental State Examination score < 17 out of 30 points).
* Severe mental disorders in the acute phase or symptomatic phase.
* Severe intellectual disability.
* Behavioural alterations as this may interfere with their participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Affect | Change from baseline affect after 90 minutes.
  The Spanish adaptation of the Positive and Negative Affect Schedule will be utilised. Participants rate how they feel at the present moment on a five-point Likert scale, where "not at all or very slightly" is scored as 1 and "a lot" as 5. Scores of two 10-item subscales will be analysed separately in the analysis, labelled either as Positive Affect or Negative Affect. Higher scores in the Positive Affect subscale represent higher levels of positive affect and lower scores in the Negative Affect subscale represent lower levels of negative affect.
Subjective Vitality | Change from baseline subjective vitality after 90 minutes.
  The 6-item Spanish adaptation of the Subjective Vitality Scale will be utilised. Participants will transmit their levels of energy and aliveness at the present moment by rating the items on a seven-point Likert scale where 1 stands for "Not true at all" and 7 "Very true". The scores for each item will be summed up for statistical analyses. Higher scores indicate higher levels of energy and aliveness feeling.

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel PÉREZ-MÁRMOL, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Granada, Faculty of Health Sciences, Granada, Spain

IPD SHARING:
Plan to Share IPD: No